CLINICAL TRIAL: NCT04589624
Title: Pilot Study of Metabolic Guidance for Therapy in Patients With Thyroid Cancer and Other Malignancies of the Head and Neck
Brief Title: An Investigational Scan (hpMRI) for Monitoring Treatment Response in Patients With Thyroid Cancer and Other Malignancies of the Head and Neck Undergoing Radiation Therapy and/or Systemic Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0482; NCI-2020-05843 (Registry Identifier: NCI-CTRP Clinical Trials Registry); 2020-0482 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-20; First posted 2020-10-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Gland Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I ( Health Volunteer MRI) (Active Comparator): Healthy volunteers undergo MRI over 30 minutes.
  Interventions: Procedure: Magnetic Resonance Imaging
- Arm II (Thyroid Cancer Patient and other malignancies of the head and neck hpMRI) (Experimental): Patients with thyroid cancer and other malignancies of the head and neck undergo hpMRI over 30 minutes at baseline, and at 1 week after the initiation of treatment. During the scan, patients also receive hyperpolarized 13-C-pyruvate IV over 30 seconds and may receive a standard MRI contrast agent at the discretion of the treating physician.
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
  Arms: Arm II (Thyroid Cancer Patient and other malignancies of the head and neck hpMRI)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
  Arms: Arm I ( Health Volunteer MRI)
Procedure: Magnetic Resonance Imaging — Undergo hpMRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
  Arms: Arm II (Thyroid Cancer Patient and other malignancies of the head and neck hpMRI)

SUMMARY:
This trial investigates whether hyperpolarized magnetic resonance imaging (hpMRI) can predict treatment response in patients with thyroid cancer and other malignancies of the head and neck undergoing radiation therapy and/or receiving systemic therapy before surgery. An hpMRI is like a standard MRI but involves the use of an imaging contrast agent called hyperpolarized 13-C-pyruvate. Diagnostic procedures, such as hpMRI, may predict a patient's response to treatment and may help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To obtain pilot metabolic imaging data from hyperpolarized magnetic resonance imaging (hpMRI) methods in patients with thyroid tumors or other malignancies of the head and neck receiving radiation therapy (XRT) and/or systemic therapy (e.g., target therapy, checkpoint inhibitors).

SECONDARY OBJECTIVE:

I. To assess early metabolic changes in response to nonsurgical therapy, including standard-of-care fractionated XRT and/or systemic therapy.

OUTLINE: Participants are assigned to 1 of 2 arms.

ARM I: Healthy volunteers undergo MRI over 30 minutes.

ARM II: Patients with thyroid cancer and other malignancies of the head and neck undergo hpMRI over 30 minutes at baseline, and at 1 week after the initiation of treatment. During the scan, patients also receive hyperpolarized 13-C-pyruvate intravenously (IV) over 30 seconds and may receive a standard MRI contrast agent at the discretion of the treating physician.

After completion of study intervention, thyroid cancer and other malignancies of the head and neck patients are followed up at 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide informed consent
* Be informed of the investigational nature of this study
* Be diagnosed with thyroid cancer and other malignancies of the head and neck with intent for treatment

Exclusion Criteria:

* Have a history of severe claustrophobia
* Have electrically, magnetically or mechanically activated implants that would preclude magnetic resonance imaging (MRI)
* Have a history of cardiac arrhythmia
* Have an allergy to Gadavist intravenous contrast
* Estimated glomerular filtration rate (eGFR) < 30
* If female, be pregnant or breast feeding at time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic imaging data from hyperpolarized magnetic resonance imaging (hpMRI) methods | 1 year
  To measure metabolic imaging data or information derived from hyperpolarized pyruvate MRI (hpMRI) that can be used to identify an early indication of response to therapy in patients with thyroid cancer. Specifically, we measure the kPL-the apparent rate constant for conversion of HP pyruvate into lactate-after one week of treatment compared to baseline measurements acquired prior to start of therapy. The kPL will be calculated from dynamic images of HP pyruvate and its metabolites. The kPL values will be calculated for each tumor and its adjacent tissue by a radiologist and physicist in conjunction using region of interest analysis to identify the margins of the tumor and surrounding normal tissue.

SECONDARY OUTCOMES:
Early metabolic changes | 1 year
  To assess early metabolic changes in response to nonsurgical therapy, including standard-of-care fractionated XRT and/or systemic therapy. The imaging biomarker for tumor metabolism, kPL, will be calculated from dynamic images of HP pyruvate and its metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Y Lai, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org